CLINICAL TRIAL: NCT03834259
Title: The Effects of Keeping the Patient in a Sitting Position for One Minute After Spinal Anesthesia on Hypotension, Nausea-vomiting and Ephedrine Consumption
Brief Title: The Effects of Keeping the Patient in a Sitting Position for One Minute After Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gulsah Karaoren, associate professor, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GK12
Record Dates: First submitted 2019-02-05; First posted 2019-02-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Hypotension; Spinal Anaesthesia
Keywords: spinal anaesthesia; ephedrine
MeSH Terms: conditions — Hypotension | interventions — Sitting Position; Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): 12.5 mg 0.5% hyperbaric bupivacaine
  Interventions: Procedure: sitting position
- Group 2 (Active Comparator): 10 mg 0.5% hyperbaric bupivacaine
  Interventions: Procedure: supine position
- Group 3 (Active Comparator): 12.5 mg 0.5% hyperbaric bupivacaine
  Interventions: Procedure: supine position

INTERVENTIONS:
Procedure: sitting position — keeping the patient in a sitting position after spinal anaesthesia
  Arms: Group 1
Procedure: supine position — keeping the patient in supine position after spinal anaesthesia
  Arms: Group 2; Group 3

SUMMARY:
The aim of this study was to examine the effect of keeping the patient in a sitting position for 1 minute after spinal anaesthesia in elective caesarean operations, primarily on the formation of hypotension and secondarily on nausea-vomiting, the need for ephedrine and the block characteristics.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 - 45 years,
* ASA physical status
* I - II,
* BMI of 25-30
* who were undergoing elective CS

Exclusion Criteria:

* vertebral anomaly,
* peripheral vascular disease,
* cardiovascular or psychiatric disorder,
* severe anemia,
* coagulopathy
* infection in the intervention region

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — the study was designed in caesarean section operations
Enrollment: 214 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
systolic arterial hypotension | every 3 minutes until the delivery and every 5 minutes until the end of surgery
  reduction of >25% in the basal systolic arterial pressure

SECONDARY OUTCOMES:
sensory block | 10 minutes after spinal block
  assesment of the time to reach T12 level with pin prick test
ephedrine requirement time | 1 hour after spinal block
  the time to first administration of ephedrine as minutes after spinal block
amount of ephedrine | 1 hour after spinal block
  administrated total ephedrine dosage as mg during surgery
surgeon and patient satisfaction | 24 hours after spinal block
  1= poor, 2=fair, 3= good, 4= very good
motor block | 24 hours after spinal block
  time to Bromage Score 0 after applying spinal block

IPD SHARING:
Plan to Share IPD: Undecided